CLINICAL TRIAL: NCT04915092
Title: Co-creation of Service Innovation - Evaluation of the Efficacy of an App for Parents to Prevent Childhood Obesity and Promote Healthy Life-styles: CoSIE Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy of an App for Parents to Promote Healthy Life-styles in Children: the CoSIE Trial
Acronym: CoSIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ID:360 - CoSIE app
Record Dates: First submitted 2020-11-16; First posted 2021-06-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-01

CONDITIONS: Childhood Obesity
Keywords: mhealth; app; obesity; prevention
MeSH Terms: conditions — Pediatric Obesity; Alzheimer Disease; Obesity

STUDY DESIGN:
Intervention Model Description: Families in the intervention arm will receive the app
Who Masked: Participant
Masking Description: Families in the control arm will receive a newsletter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The app is explained and installed during the recruitment to the family in the intervention group. Some families in this group will be selected to take part to the qualitative research.
  Interventions: Device: CoSIE app
- Control group (No Intervention): Every months during the first year of study a newsletter is sent only to the members of the control group.

INTERVENTIONS:
Device: CoSIE app — The app is a mobile phone application compatible with both iOS and Android operating system. Parents are able to register their children and to keep track of their weight status and activities. The app include five themes: child development, physical activity, healthy food, critical situations, BMI.
  Push notification on healthy behaviours, on important event taking place in the province of Reggio Emilia, on food advices based on seasonality and on party tips are constantly delivered by the app.
  Arms: Intervention group

SUMMARY:
The objective of the study is to evaluate the effectiveness of the app in terms of changing lifestyles both related to nutrition and physical activity. The study is also aimed at evaluating the usability and the degree of acceptance of the app among parents.

The primary objective will be assessed in terms of the change in the consumption of sugary drinks and high-calorie food and in terms of time spent in front of a screen.

The secondary objectives are the evaluation of BMI (percentile and z-score) and waist circumference and the evaluation of the usability of the app.

STUDY DESIGN The study is a randomized control trial. Both parents and children are recruited.

* Family paediatricians during the health balance of 3 or 5 years old (children between 3 and 6.5 years old)
* Sport medicine during the visits for sport ability (children between 7 and 11 years old)
* Pediatric Endocrinology and Diabetology of the Santa Maria Hospital during routine visits (children between 5 and 11 years old)

When the study is presented to families, few clinical information are collected on the electronic platform designed for enrollment and randomization:

* Child weight and height
* Child waist circumference

More information about children and parents are collected (through questionnaire).

The families (both treatment and control ) are contacted after 12 month and after 24 months from the recruitment to answer to a questionnaire on lifestyle habits (food and physical activity) of the child and app utilization

During this visit also child weight, height and waist circumference will be collected.

Intervention group The app is explained and installed during the recruitment to the family in the intervention group.

Some families in this group will be selected to take part to the qualitative research.

Control group Every months during the first year of study a newsletter is sent only to the members of the control group.

DETAILED DESCRIPTION:
Childhood obesity is a highly prevalent condition and together with the behaviours associated with it, such as improper diet and physical inactivity, it generates a high burden of disease in adulthood.

In recent years, it is increasing the use of mobile devices in support of health prevention and promotion strategies. In a primary care setting these new technologies offer the opportunity to open a two-way communication channel between parents and institutions and can help by adapting the intervention and framing the message according to the needs of each family.

Since 2010, the Reggio Emilia AUSL has started a research and interventions program aimed at preventing childhood obesity. The program has adopted a multilevel and multi-setting strategy for primary prevention (BMInforma Program).

Since 2017, together with the University of Bologna and the regional company Lepida2000, the Local Health Authority is part of the Co-creation of Service Innovation in Europe project (CoSIE Project), a project funded by the European Union with a Horizon 2020 call coordinated by the University of Turku, Finland. The CoSIE project promotes the co-creation of public services through the involvement of citizens and other interested parties in the definition of objectives and delivery methods.

The project is divided into nine pilot projects and the Italian pilot project, carried out in the province of Reggio Emilia, is part of the AUSL program for the prevention of childhood obesity. The aim of the pilot project is to create a network between the services involved in the prevention and treatment of obesity and, at the same time, it aims to create an app that can help promote a healthy lifestyle. The app was designed and created with a co-creation process.

The objective of the study is to evaluate the effectiveness of the app in terms of changing lifestyles both related to nutrition and physical activity. Furthermore,an aim of the study is to evaluate the usability and the degree of acceptance of the app among parents.

The primary objective will be assessed in terms of the change in the consumption of sugary drinks and high-calorie food and in terms of time spent in front of a screen.

The secondary objectives are the evaluation of BMI (percentile and z-score) and waist circumference and the evaluation of the usability of the app.

STUDY DESIGN The study is a randomized control trial.

Both parents and children are recruited. The recruitment is done by some members of the CoSIE project Consulting Committee:

* Family paediatricians during the health balance of 3 or 5 years old (children between 3 and 6.5 years old)
* Sport medicine during the visits for sport ability (children between 7 and 11 years old)
* Pediatric Endocrinology and Diabetology of the Santa Maria Hospital during routine visits (children between 5 and 11 years old)

When the study is presented to families, few clinical information are collected on the electronic platform designed for enrollment and randomization:

* Child weight and height
* Child waist circumference

More information about children and parents are collected (through questionnaire).

The families (both treatment and control ) are contacted after 12 month and after 24 months from the recruitment to answer to a questionnaire on lifestyle habits (food and physical activity) of the child and app utilization

During this visit also child weight, height and waist circumference will be collected.

Intervention group The app is explained and installed during the recruitment to the family in the intervention group.

Some families in this group will be selected to take part to the qualitative research.

Control group Every months during the first year of study a newsletter is sent only to the members of the control group.

ELIGIBILITY:
Inclusion Criteria:

* parents of children aged 3 to 11 presneting for a new well child visit or for a sport medicin visit or presenting for a childhood obesity visit at the AUSL Reggio Emilia clinics, including family pediatricians clinics.

Exclusion Criteria:

* Families resident outside the Province of Reggio Emilia
* Parents with no comprehension of the Italian language
* Children inside a program for obesity cure or prevention. The program are:

  * the GET program (a program coordinated by the hospital pediatric unit in which obese children follow a group intervention),
  * the BMInforma program (in which overweight girls from 5 to 7 years old follow a counselling proposed by the family paediatrician),
  * the second level medical clinic in which obese children with pathologic condition are cured
* Children with severe obesity previously diagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in consumption of sugar - sweetened beverages and juice, first year | 12 months
  Endpoint: number per week Outcome: Delta 12m-baseline Test/analysis: Difference between groups Source: Questionnaire in FU visits
Change in consumption of sugar - sweetened beverages and juice, second year | 24 months
  Endpoint: number per week Outcome: Delta 24m - baseline Test/analysis: Difference between groups Source: Questionnaire in FU visits
Change in consumption of hypercaloric foods like fried food, salty snacks and sweet snacks/candies, first year | 12 months
  Endpoint: number per week Outcome: Delta 12m-baseline Test/analysis: Difference between groups Source: Questionnaire in FU visits
Change of consumption of hypercaloric foods like fried food, salty snacks and sweet snacks/candies, second year | 24 months
  Endpoint: number per week Outcome: Delta 24m-baseline Test/analysis: Difference between groups Source: Questionnaire in FU visits
Change in screen time spent by children, first year | 12 months
  Endpoint: Minutes of screen time per day Outcome: Delta 12m-baseline Test/analysis: Difference between groups Source: Questionnaire in FU visits
Change in screen time spent by children, second year | 24 months
  Endpoint: Minutes of screen time per day Outcome: Delta 24m-baseline Test/analysis: Difference between groups Source: Questionnaire in FU visits

SECONDARY OUTCOMES:
BMI centile of children after the first year | 12 months
  Endpoint: BMI centile Outcome: Delta 12m-baseline Test/analysis: Difference between group means Source: FU visits
BMI centile of children after the second year | 24 months
  Endpoint: BMI centile Outcome: Delta 24m-baseline Test/analysis: Difference between group means Source: FU visits
Acceptability | after at 12 months of app utilization
  How much parents accept the concept of using an app to guide their habits in children education Test/analysis: qualitative analysis Source: Interviews
Usability | after at 12 months of app utilization
  How much each single app function is used and is perceived as useful by parents Test/analysis: qualitative analysis Source: Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Giorgi Rossi, phd, Principal Investigator — Azienda USL-IRCCS Reggio Emilia
Locations (1):
- Azienda USL-IRCCS Reggio Emilia, Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giorgi Rossi P, Ferrari F, Amarri S, Bassi A, Bonvicini L, Dall'Aglio L, Della Giustina C, Fabbri A, Ferrari AM, Ferrari E, Fontana M, Foracchia M, Gallelli T, Ganugi G, Ilari B, Lo Scocco S, Maestri G, Moretti V, Panza C, Pinotti M, Prandini R, Storani S, Street ME, Tamelli M, Trowbridge H, Venturelli F, Volta A, Davoli AM; Childhood Obesity Prevention Working Group. Describing the Process and Tools Adopted to Cocreate a Smartphone App for Obesity Prevention in Childhood: Mixed Method Study. JMIR Mhealth Uhealth. 2020 Jun 8;8(6):e16165. doi: 10.2196/16165. PMID 32357123